CLINICAL TRIAL: NCT05636488
Title: Determination of the Effects of Noise Level in the Operating Room on the Anesthesiologist, Patient, and Environment During the Induction Phase and Investigation of the Effect of Staff Training
Brief Title: Determination of the Effects of Noise Level in the Operating Room
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Begüm Nemika Gökdemir, Research Assistant, Baskent University
Other Study IDs: 2022-07/1932
Record Dates: First submitted 2022-11-13; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Noise; Adverse Effect; Noise Induced Hearing Loss
Keywords: noise induced hearing loss; operatin room's noise
MeSH Terms: conditions — Hearing Loss, Noise-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — There is no intervention group in this study

SUMMARY:
The goal of this observational study is to learn about effects of noise in healthy patients undergoing elective surgery.

DETAILED DESCRIPTION:
There are many factors that can negatively affect surgical performance in operating rooms. Noise is the most striking of these factors. Excessive noise can cause hearing loss, cognitive dysfunction, anxiety, stress-induced increases in cortisol levels, and an increased risk of cardiovascular disease. Noise can have negative effects on concentration and performance. At the same time, workplace noise is one of the most important causes of fatigue. One of the anesthesia phases where the sound level reaches the highest levels is the induction phase. With this study, the investigators want to examine the effects on the anesthesia team, the patient and the environment by measuring the noise levels during the induction period, and then train the operating room personnel to examine the effects on this issue. The investigators aim to raise awareness about the development of procedures and training programs for operating room personnel.

ELIGIBILITY:
Inclusion Criteria:

* patients over the age of 18,

  * Elective cases to be taken under general anesthesia,
  * Those who do not have a psychiatric disease,
  * Patients without hearing loss

Exclusion Criteria:

* patients under the age of 18
* Patients who have psychiatric disease
* Patients who has hearing loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 without hearing loss who will undergo elective surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
assessing effect of noise level on fatigue with questionnaire | postoperative 24 hours
  A quieter environment can be created if noise level can be shown to cause fatigue in work performance.
assessing effect of noise level on anxiety with questionnaire | postoperative 24 hours
  A quieter environment can be created if noise level can be shown to cause anxiety in work performance.

IPD SHARING:
Plan to Share IPD: No